CLINICAL TRIAL: NCT06132724
Title: Observation et Mise en Relation Des Transitions Cardio-respiratoires et Motrices à la frontière de l'Exercice modéré
Brief Title: Observation and Interactions Between Cardio-respiratory and Motor Transitions at the Limits of Moderate Exercise.
Acronym: CAREMO
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: TIMC-IMAG (Other); University Grenoble Alps (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC23.0263
Record Dates: First submitted 2023-11-09; First posted 2023-11-15 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Healthy
Keywords: Retraining; Physical Activity; First Ventilatory Threshold; Moderate Intensity Domain; Physiological Transitions; Motricity; Cardiorespiratory; Connected Objects
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Volunteers: Subjects who will agree to participate to the study will be healthy subject with no particular antecedents.
  Subjects will be enroled for two sessions with a 20 min monitoring phase in each session, to coect physiological data with non invasive sensors.
  Interventions: Other: Signal acquisition

INTERVENTIONS:
Other: Signal acquisition — Synchronized signals from cardiac, respiratory and movements non invasive measurements.
  One acquisition is 20 minutes long, and each subject participate to two sessions, separated by 1 to 15 days.

SUMMARY:
The goal of this observational study is to learn about physiological transitions around the limit of moderate exercise intensity on cardiac, respiratory and motor modalities, in healthy population.

The main questions it aims to answer is:

* is it possible to define criteria on cardiac, respiratory and motor modalities to identify transitions?
* are those transitions visible on embedded and non-intrusive monitoring equipment?
* are those identified transitions somehow connected to first ventilatory threshold (VT1)?

Participants will do a sub-maximal effort test on cycloergometer calibrated to make them cross their first ventilatory threshold.

DETAILED DESCRIPTION:
Cycling is a commonly prescribed activity when it comes to physical activities for rehabilitation. Because it is soft and progressive effort, cycling suits well for patients with chronic conditions (diabete, cancer, fibromyalgia, ...) For safety and effectiveness of the activity, it is necessary to prescribe activity at a regular and moderate intensity. This can be achieved by personalizing intensities to match specifically the patient health condition in order to build an efficient and progressive rehabilitation program.

Physical activity prescription rely on four pillars: frequency, duration, volume and intensity. While first three pillars are quite easy to regulate,effort intensity is harder to handle on training planning. It is harder to measure, and defining personalized guideline for practice is more complex.

It is known that first ventilatory threshold (VT1) is a individualized marker representing the higher limit of moderate intensity effort zone. It makes it an interesting tool for the prescription of intensity for retraining purposes: it guaranties a safe practice, intense enough to make beneficial physiological adaptations for the patient.

In this retraining context and with this study, we aim to identify markers of this transition on cardiac, respiratory and motor modalities, with embedded and non intrusive equipment, during a sub-maximal effort test in laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Capability to cycle during 20min
* No contraindication to cycling at a moderate pace
* No acute pathology (less than 2 years old)
* No cardiac or respiratory chronic pathology
* No locomotive problem on the spine or the lower limbs
* No recent injuries (less than 2 months)
* Stature compatible with the use of the plethysmography t-shirt

Exclusion Criteria:

* Pregnant (urine strip test) or breastfeeding women
* Persons referred to in articles L1121-5 to L1121-8 of the CSP (protected persons) person deprived of liberty by judicial or administrative decision, person subject to a legal protection measure
* Subject being excluded from another study
* Subject who reached the ceiling of 4500 euros due to their participation in other studies involving human in the past 12 months

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Heathy volunteers with various physical conditions
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-12-05 (Actual); Primary Completion 2024-06-11 (Actual); Study Completion 2024-06-11 (Actual)

PRIMARY OUTCOMES:
Database of physiological signals | 20 minutes
  Synchronized signals from embedded and non-intrusive connected devices for cardiorespiratory and motricity measurements and equivalent laboratory measurements during cycling on a cyclo-ergometer

SECONDARY OUTCOMES:
Evaluation of the feeling of wearing equipment | 15 minutes
  Questionnaire at the end of each session to assess the comfort / discomfort wearing the equipment used during the test
Criteria for the observation of a respiratory transition | 6 months
  Feasibility of the transition detection, repeatability of the detection with the respiratory criteria
Criteria for the observation of a cardiac transition | 6 months
  Feasibility of the transition detection, repeatability of the detection with the cardiac criteria
Criteria for the observation of a motricity transition | 6 months
  Feasibility of the transition detection, repeatability of the detection with the motricity criteria
Multi-modal prediction of the first ventilatory threshold | 6 months
  Correlation with the measurement of ventilatory threshold 1 (VT1)

CONTACTS AND LOCATIONS:
Locations (1):
- Plateforme PRETA P3I, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blair SN. Physical inactivity: the biggest public health problem of the 21st century. Br J Sports Med. 2009 Jan;43(1):1-2. No abstract available. PMID 19136507
- [Background] Pisot R. Physical Inactivity - the Human Health's Greatest Enemy. Zdr Varst. 2021 Dec 27;61(1):1-5. doi: 10.2478/sjph-2022-0002. eCollection 2022 Mar. PMID 35111260
- [Background] Meyler S, Bottoms L, Muniz-Pumares D. Biological and methodological factors affecting V̇O2max response variability to endurance training and the influence of exercise intensity prescription. Exp Physiol. 2021 Jul;106(7):1410-1424. doi: 10.1113/EP089565. Epub 2021 Jun 8. PMID 34036650
- [Background] Succi PJ, Dinyer TK, Byrd MT, Bergstrom HC. Comparisons of the Metabolic Intensities at Heart Rate, Gas Exchange, and Ventilatory Thresholds. Int J Exerc Sci. 2020 May 1;13(2):455-469. doi: 10.70252/IBRC8606. eCollection 2020. PMID 32509109
- [Background] Pouliquen C, Nicolas G, Bideau B, Garo G, Megret A, Delamarche P, Bideau N. Spatiotemporal analysis of 3D kinematic asymmetry in professional cycling during an incremental test to exhaustion. J Sports Sci. 2018 Oct;36(19):2155-2163. doi: 10.1080/02640414.2018.1432066. Epub 2018 Jan 30. PMID 29381424
- [Background] Jamnick NA, Pettitt RW, Granata C, Pyne DB, Bishop DJ. An Examination and Critique of Current Methods to Determine Exercise Intensity. Sports Med. 2020 Oct;50(10):1729-1756. doi: 10.1007/s40279-020-01322-8. PMID 32729096